CLINICAL TRIAL: NCT07212244
Title: A Prospective, Long-term Analysis of Clinical Outcomes in Patients Undergoing Magnetic Resonance-Guided Focused Ultrasound for Medication-Refractory Tremor
Brief Title: Analysis of Clinical Outcomes in Patients Undergoing Magnetic Resonance-Guided Focused Ultrasound for Medication-Refractory Tremor
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Other Study IDs: 6830
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Essential Tremor; Essential Tremor, Movement Disorders
Keywords: Focused Ultrasound; Thalamotomy; Hand tremor; MRI-guided focused ultrasound (MRgFUS); Primidone; Propranolol
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Magnetic Resonance-Guided Focused Ultrasound (MRgFUS) Thalamotomy: Patients with medication-refractory essential tremor who are scheduled to undergo MRgFUS thalamotomy at Sunnybrook Health Sciences Centre as part of standard of care. Eligible participants providing informed consent will be enrolled and followed prospectively for a minimum of 3 years to evaluate long-term efficacy and safety outcomes.

SUMMARY:
The goal of this observational study is to evaluate the long-term efficacy and safety of MR-guided focused ultrasound (MRgFUS) thalamotomy in patients with medication-refractory essential tremor.

The main questions it aims to answer are:

1. Does MRgFUS thalamotomy provide sustained reduction in tremor severity over 3 years?
2. What are the long-term neurological and quality-of-life outcomes associated with this procedure?

Participants will:

* Undergo MRgFUS thalamotomy as part of standard of care at Sunnybrook Health Sciences Centre.
* Be followed prospectively for a minimum of 3 years with scheduled assessments including:

  1. Clinical Rating Scale for Tremor (CRST)
  2. Neurological exams and adverse event monitoring
  3. Quality of Life in Essential Tremor (QUEST) questionnaire
  4. Scale for the Assessment and Rating of Ataxia (SARA)
  5. MRI imaging and neuropsychological testing

DETAILED DESCRIPTION:
This single-centre, prospective observational cohort study will evaluate long-term outcomes of MR-guided focused ultrasound (MRgFUS) thalamotomy for medication-refractory essential tremor at Sunnybrook Health Sciences Centre. It is anticipated that about 240 people will be recruited into this study over the next 6 years. It is expected that this study will take 6 years to complete and that results will be known in 6-7 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22 years or older
2. Able and willing to give consent and to attend all visits
3. Diagnosed with essential tremor that is refractory to at least two first-line tremor medications
4. Confirmed to have moderate-to-severe hand tremor by the MRI guided Focused Ultrasound (MRgFUS) neurology team
5. Deemed suitable surgical candidates (decision-to-treat) by the MRgFUS neurosurgical team

Exclusion Criteria:

1. Patients with standard contraindications to MRI such as non-MRI compatible implants or devices
2. Patients deemed clinically unfit to undergo MRgFUS thalamotomy due to health status including (but not limited to) pregnancy, advanced kidney disease, unstable cardiac status, severe hypertension, cerebrovascular disease, brain tumour, pulmonary disorders
3. Receiving anti-coagulants or drugs known to increase risk of hemorrhage within 2 weeks of MRgFUS procedure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 22 years and older with medication-refractory essential tremor and moderate-to-severe hand tremor who are scheduled to undergo MR-guided focused ultrasound (MRgFUS) thalamotomy at Sunnybrook Health Sciences Centre as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2031-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Change in tremor severity measured by Clinical Rating Scale for Tremor (CRST) | Assessments occur at baseline; Day 1; Week 12; and at 1, 2, and 3-year follow-up visits post-treatment.
  CRST is a validated scale assessing tremor severity through clinical examination and functional tasks. Tremor scores range from 0 (no tremor) to 32 for the dominant hand and 0 to 28 for the non-dominant hand, with higher scores indicating greater tremor severity. Change from baseline will be assessed. CRST measures will be videotaped following a standardized script.

SECONDARY OUTCOMES:
Standardized Neurological Examination and Adverse Events (AEs) | Assessments occur at baseline; Day 1; Week 12; and at 1, 2, and 3-year follow-up visits post-treatment.
  Adverse events will be recorded and graded according to CTCAE v5.0. AEs will be recorded and categorized according to severity, and relationship to procedure.
Quality of Life in Essential Tremor (QUEST) questionnaire | Assessments occur at baseline; Week 12; and at 1, 2, and 3-year follow-up visits post-treatment.
  The QUEST is a self-reported, validated survey scoring the physical, psychosocial, communication, hobbies/leisure and work/finance domains of the life of a patient with Essential Tremor. Participants rate their level of agreeance with 30 statements on a 5-point scale (0 to 4), for a maximum score of 120. Higher scores reflect poorer quality of life.
Scale for the Assessment and Rating of Ataxia (SARA) | Assessments occur at baseline; Day 1; Week 12; and at 1, 2, and 3-year follow-up visits post-treatment.
  The SARA is a validated, comprehensive ataxia scale, and comprises 8 items carrying a maximum total score of 40 points. Higher scores suggest increased ataxia. The SARA will be used to compare degree of ataxia between baseline and the follow-up visits. In particular, the SARA will be used to assess changes in gait and stance associated with the procedure.
Change in MRI Measures | Assessments occur at baseline; Day 1; Week 12; and at 1-, 2-, and 3-year follow-up visits post-treatment.
  MRI sequences (T1, T2*, DTI, resting state fMRI) will be obtained to assess treatment-related changes and safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No